CLINICAL TRIAL: NCT00571545
Title: The Effect of Exercise on Mood After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kathleen Bell, Professor, Department of Rehabilitative Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22868-B; H133A020508
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Traumatic Brain Injury; Depression
Keywords: Traumatic brain injury; Depression; Exercise
MeSH Terms: conditions — Brain Injuries, Traumatic; Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects recruited from the community with a history of traumatic brain injury were enrolled into a 10 week supervised exercise program and encouraged to exercise at home as well.
  Interventions: Behavioral: Aerobic exercise
- 2 (Other): Controls were wait-listed for the supervised exercise program but were not treated during the 10 week wait period.
  Interventions: Behavioral: No exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — A supervised aerobic exercise program occurred weekly for 30 minutes with a 15 minute warm-up and a 15 minute cool down. A half hour educational session on aspects of exercise and overcoming barriers to exercise was also instituted.
  Arms: 1
Behavioral: No exercise — Controls were wait-listed for the exercise program during the 10 week study period.
  Arms: 2

SUMMARY:
We proposed to examine the effect of an aerobic exercise intervention on depression in persons with Traumatic Brain Injury (TBI). We will compare persons with chronic brain injury who are assigned to receive the exercise intervention with those in the control group to determine the effect of exercise on levels of depression and specific symptoms related to depression including anxiety, pain, sleep, and cognition. In addition, the effect of exercise on activity, participation level, and quality of life will be examined.

HYPOTHESES:

1. Participation in an aerobic exercise intervention will decrease the severity of depression in persons with chronic TBI.
2. Participation in an aerobic exercise intervention will lead to improvements in negative symptoms associated with depression including anxiety, insomnia, pain, and impaired cognitive functioning.
3. Participation in an aerobic exercise intervention will be related to improvements in activity and participation for patients with TBI.
4. Participation in an aerobic exercise intervention will lead to improvements in perceptions of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury 1-5 years prior to enrollment
* Current depression as measured by a score of 5 or greater on the depression portion of the Physician Health Questionnaire (PHQ).
* Sufficient cognitive ability to maintain participation in the study
* Sufficient English language ability to allow participation without an interpreter

Exclusion Criteria:

* Current suicidal ideation with intent or plan
* Currently pregnant
* History of significant cardiovascular or respiratory disease
* History of significant cardiovascular or respiratory disease
* Physical barriers to the use of standard aerobic exercise equipment

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2004-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 10 week

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Bell, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Hoffman JM, Bell KR, Powell JM, Behr J, Dunn EC, Dikmen S, Bombardier CH. A randomized controlled trial of exercise to improve mood after traumatic brain injury. PM R. 2010 Oct;2(10):911-9. doi: 10.1016/j.pmrj.2010.06.008. PMID 20970760